CLINICAL TRIAL: NCT06504823
Title: The Effect of Light Level Applied During Breastfeeding on Maternal Stress, Anxiety, Psychological Well-being and Breastfeeding Motivation Randomize Plasebo kontrollü çalışma
Brief Title: The Effect of Light Level Applied During Breastfeeding on Maternal Stress, Anxiety, Psychological Well-being and Breastfeeding Motivation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emine Yıldırım (Other)
Responsible Party: Sponsor-Investigator, Emine Yıldırım, Assistant Professor, Osmaniye Korkut Ata University
Organization: Osmaniye Korkut Ata University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1111112
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Stress; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo group (Placebo Comparator)
  Interventions: Other: Light level
- experimental group (Experimental)
  Interventions: Other: Light level

INTERVENTIONS:
Other: Light level — light application

SUMMARY:
To determine the effect of the light level applied during breastfeeding on the mother's stress, anxiety, psychological well-being and breastfeeding motivation. This research was planned as a single-blind randomized controlled experimental type study comparing separate groups as intervention-placebo controlled. Data will be collected with the Introductory Information Form, Psychological Well-Being Scale, Perceived Stress Scale (ASÖ/PSÖ-14), State-Trait Anxiety Inventory (STAI) and Breastfeeding Motivation Scale (For Primiparous Mothers). The effect of two different light levels on mothers will be examined.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years of age or older, volunteering.

Exclusion Criteria:

* Having any problem that prevents communication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-22 (Estimated); Primary Completion 2024-07-26 (Estimated); Study Completion 2024-08-02 (Estimated)

PRIMARY OUTCOMES:
stress | 1 day
  stress scale

SECONDARY OUTCOMES:
anxiety | 1 day
  anxiety scale